CLINICAL TRIAL: NCT05667805
Title: Coagulation in Cirrhosis
Acronym: COUCH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, PhD, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1144/2022
Record Dates: First submitted 2022-12-16; First posted 2022-12-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Liver Cirrhosis
Keywords: Patient Blood Management; Platelet Concentrates; Transfusion; Coagulation
MeSH Terms: conditions — Liver Cirrhosis; Thrombosis | interventions — Factor IX; prothrombin complex concentrates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: interventional radiologists
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal substitution of human prothrombin complex and/or platelet concentrates (Active Comparator): If INR < 1,5: 10 I.E. human prothrombin complex/kg bodyweigt/0,5 INR AND/OR If platelets < 50 G/l: ((50 G/l - measured thrombocyte concentration G/l) x total blood volume) platelet concentrate
  Interventions: Drug: Platelet Concentrate; Drug: Prothrombin Complex Concentrate
- Restrictive substitution of human prothrombin complex and/or thrombocytes (Experimental): No substitution of blood products described in the Active Comparator group.
  Interventions: Other: Restricitve Use

INTERVENTIONS:
Drug: Platelet Concentrate — Liberal use (standard treatment)
  Arms: Liberal substitution of human prothrombin complex and/or platelet concentrates
Drug: Prothrombin Complex Concentrate — Liberal use (standard treatment)
  Other Names: PPSB
  Arms: Liberal substitution of human prothrombin complex and/or platelet concentrates
Other: Restricitve Use — Restrictive use of human prothrombin complex and platelet concentrates. No prophylactic substitution.
  Arms: Restrictive substitution of human prothrombin complex and/or thrombocytes

SUMMARY:
Out of fear of bleeding, liver cirrhosis patients are often treated prophylactically with blood and coagulation products before minor interventions. The COUCH study will examine whether these patients benefit from a restrictive administration of coagulation products.

DETAILED DESCRIPTION:
Patients with cirrhosis commonly have deranged coagulation parameters, in particular thrombocytopenia and/or an increased INR. However, these laboratory findings do not necessarily correlate with an increased tendency of bleeding. In fact, the reduced synthesis of both pro- and anticoagulant factors often equates to a new equilibrium in the coagulation system. Nevertheless, out of fear of bleeding, liver cirrhosis patients with deviated laboratory coagulation parameters are often aggressively treated with coagulation products (such as platelet concentrates and prothrombin complex concentrate (PCC)) before minor interventions and punctures. Since these products can also have procoagulant side effects, we will investigate whether patients with liver cirrhosis without a history of bleeding or clinical bleeding signs benefit from a restrictive substitution regime. The study will be carried out monocentrically at the General Hospital of Vienna, and will include 400 patients divided into two groups (liberal vs. restrictive substitution of thrombocytes and/or PCC) over an est. period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

Patients at the University Hospital of Vienna with diagnosed liver cirrhosis and deranged coagulation parameters (INR >1,5 AND/ OR platelet count <50 G/L) who are scheduled for one of the following elective invasive interventions of the liver

* Biopsy or puncture
* Microwave ablation (MWA) or radiofrequency ablation (RFA)
* Transjugular intrahepatic portosystemic shunt (TIPS)
* Percutaneous transhepatic cholangiography drain (PTCD)

Exclusion Criteria:

* Missing informed consent or inability to consent
* Age < 18 years
* Pregnancy or breastfeeding
* Manifest ascites
* Chronic kidney injury stage G4 or G5, KDIGO
* Uninterrupted anticoagulant therapy, except for acetylsalicylic acid (ASA)
* History of bleeding or clinical signs of a hemorrhagic diathesis in the physical examination (e.g., petechia, ecchymosis, mucosal bleeding, hemorrhagic diathesis within the family, menorrhagia, prolonged bleeding after surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Major Bleeding | 3 days
  bleeding complication within 3 days after the intervention

SECONDARY OUTCOMES:
bleeding complication | 28 days
  bleeding complication within 28 days after the intervention
thromboembolic events | 28 days
transfusion related complications | 28 days
28 day overall mortality | 28 days
28 day bleeding related mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of the Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided